CLINICAL TRIAL: NCT04324710
Title: Peripheral Gene Expression of Endocannabinoid System Components in Episodic and Chronic Migraine Patients: a Pilot Study
Brief Title: Gene Expression of Endocannabinoid System in Episodic and Chronic Migraine Patients
Status: Completed | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: ES2020
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Chronic Migraine
Keywords: Endocannabinoids; Medication overuse; Peripheral blood mononuclear cells
MeSH Terms: conditions — Prescription Drug Overuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Since PBMCs contain the full complement of epigenetic enzymes found in most tissues, the investigators evaluated the role of DNA methylation in the regulation of ES gene transcription in all the enrolled subjects.
  DNA was extracted from whole blood using QIAmp DNA Blood Mini Kit and its concentration was determined by NanoDrop quantification. Arrays preparation and data analysis were performed by Genomix4Life srl. High-quality DNA (500 ng) was bisulfite converted using EZ DNA methylation kit. Bisulfite converted DNA (200ng) was used for analysis of whole-genome methylation, using the HumanMethylation 450 K BeadChip, which contains 485 577 probes covering 21 231 (99%) RefSeq genes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preclinical and clinical evidence suggests a role for the dysregulation of endocannabinoid system (ES) in migraine pain, particularly in subjects with chronic migraine.

The gene expression of ES components were assayed in peripheral blood mononuclear cells (PBMCs) of patients with episodic migraine (EM), chronic migraine with medication overuse (CM-MO) and age-matched healthy controls (CT). It was evaluated the protein expression of cannabinoid receptors (CB) 1 and 2 as well as DNA methylation changes in genes involved in ES components.

DETAILED DESCRIPTION:
Migraine is a neurovascular disease whose pathophysiology is far from being completely clarified. This is mainly due to the complex mechanisms that underlie migraine attack as well as its recurrence. The endocannabinoid system (ES) is a complex signalling system involved in different biological processes (e.g. neuronal activity, pain sensation and immune functions) and it plays a crucial role in the maintenance of body homeostasis. The ES components include the endogenous lipids, the most studied ones being N-arachidonoylethanolamide (AEA) and 2-arachidonoylglycerol (2-AG), their metabolic enzymes and at least two cannabinoid receptors (CB1 and CB2). The biosynthesis of AEA mainly occurs by N-acylphosphatidylethanolamide-phospholipase D (NAPE-PLD), whereas 2-AG is produced through the action of diacylglycerol lipase (DAGL). AEA is metabolized by fatty acid amide hydrolase (FAAH) and 2-AG mainly by monoacylglycerol lipase (MAGL).

Alterations in gene expression of ES components may involve various cell types, multiple catabolic pathways and the generation of active metabolites via epigenetic mechanisms, under both physiological and pathological conditions. CB genes, for instance, may interact with different transcriptional factors, many of which are related to DNA methylation and histone post-translational modifications. A dysfunctional ES has been associated to numerous disorders including migraine. The ES, indeed, modulates multiple activities and neuromodulators/neurotransmitters that play a crucial role in migraine pathogenesis. ES is also implicated in the descending modulation of the trigeminovascular nociceptive transmission from the brainstem afferents. Previous studies from the Laboratory of Neurophysiology of Integrative Autonomic Systems, Headache Science Centre, IRCCS Mondino Foundation, Pavia (Italy), using the migraine-specific animal model based on nitroglycerin administration in rat, demonstrated the existence of interactions between the ES and pain mediation. In particular, the investigators showed a key role for AEA and for FAAH-regulated AEA activity in the processing of trigeminal nociceptive signals. AEA inhibits neurogenic dural vasodilatation, as well as calcitonin gene-related peptide-induced and nitric oxide-induced dural vessel dilation, an activity that is reversed by CB1 antagonism. The interaction between the ES and migraine pain is also suggested by clinical observations. FAAH activity was higher in platelets of women with episodic migraine (EM) to suggest a more marked degradation of AEA. Subjects with chronic migraine (CM) and medication overuse (MO) showed an altered endocannabinoid metabolism not only in platelets, but also in the CSF. Although the above clinical findings are scattered and replicated, their re-consideration in the light of more recent data from the increasing pre-clinical evidence prompt the need to investigate in more depth the role of ES in migraine pathophysiology.

Several studies suggest that changes in ES components detected in peripheral blood mononuclear cells (PBMCs) are reliable indicators of a central dysfunction of the ES in different neurological diseases. For instance, in patients with Parkinson disease or multiple sclerosis, increased CSF levels of AEA were associated with a reduction in the activity and protein content of FAAH in PBMCs, which is indicative of an increased AEA tone. AEA levels were elevated in the CSF and in the blood of schizophrenic subjects, with a significant drop in AEA blood levels and in mRNA transcripts of CB2 and FAAH in PBMCs following clinical remission.

The aim of this study, was the identification of specific functional patterns of ES activity in subjects with migraine. To this end, the investigators performed a thorough evaluation of multiple peripheral components of the ES (gene expression, protein expression and DNA methylation) in PBMCs of representative samples of subjects with EM without aura, CM-MO and in healthy controls (CT).

Twenty-five subjects with EM, 26 with CM-MO and 24 CT were enrolled in the headache center of the IRCCS Mondino Foundation of Pavia (Italy). The study was approved by the local Ethics Committee and all subjects enrolled signed a written informed consent.

Blood samples (20ml) were collected within ethylenediamine tetra-acetic acid (EDTA) containing tubes from participants. Blood samples were diluted in 1:1 ratio with phosphate buffer saline 1X (PBS 1X) (Sigma). Diluted blood samples were slowly loaded onto Ficoll separating solution (15ml) (Sigma) and centrifuged at 800 g without brake for 30 min at room temperature. PBMCs accumulated as the middle white monolayer, were washed twice in sterile PBS 1X and centrifuged at 300 g for 15 min. For each sample, a batch of PBMCs was used for RNA or DNA extraction and another one for flow-cytometer analysis.

In the PBMCs isolated from the subjects in the 3 study groups the investigators assayed:

* CB1 and CB2 protein expression;
* expression of the following genes: CB receptors, FAAH, NAPE-PLD, MAGL and DAGL
* DNA methylation of ES components. To determine the relative level of CB1 and CB2 protein expression in PBMCs, the investigators used flow-cytometry with a FACS Canto flow-cytometer (Becton-Dickenson). After isolation, cells (100000 per reaction) were stained using antibodies against CD45 (BD Biosciences, 1:50), CB1 (R&D system, 1:50) and CB2 receptors (Cayman Chemical, 1:30); a total of 10000 events were counted in windows gated for the intersection of CD45 staining with CB1 and CB2.

Total RNA from PBMCs was isolated using standard procedure (Zymo Research) and RNA quality was assessed using a nanodrop spectrophotometer (Nanodrop™ Thermo Fisher Scientific); cDNA was generated using the iScript cDNA Synthesis kit (Biorad) following the supplier's instructions. Gene expression of CB receptors, FAAH, NAPE-PLD, MAGL and DAGL was analyzed using the Fast Eva Green supermix (BIO-RAD). Ubiquitin (UBC), whose expression remained constant in all experimental groups, was used as housekeeping gene. The amplification was performed with a light Cycler 480 Instrument rt-PCR Detection System (Roche) following the supplier's instructions. All samples were assayed in triplicate and gene expression levels were calculated according to 2-∆Ct = 2- (Ct gene - Ct housekeeping gene) formula by using Ct values.

Since PBMCs contain the full complement of epigenetic enzymes found in most tissues, including neurons and peripheral nucleated cells, the investigators evaluated the role of DNA methylation in the regulation of ES gene transcription in all the enrolled subjects.

DNA was extracted from whole blood using QIAmp DNA Blood Mini Kit (Qiagen) and its concentration was determined by NanoDrop quantification (NanoDrop Techologies, Thermofisher). Arrays preparation and data analysis were performed by Genomix4Life srl (Baronissi, Italy). High-quality DNA (500 ng) was bisulfite converted using EZ DNA methylation kit (Zymo Research, Irvine, CA, USA). Bisulfite converted DNA (200ng) was used for analysis of whole-genome methylation, using the HumanMethylation 450 K BeadChip (Illumina, San Diego, CA, USA), which contains 485 577 probes covering 21 231 (99%) RefSeq genes. In brief, bisulfite converted DNA was whole-genome amplified for 20 h followed by end-point fragmentation. Fragmented DNA was precipitated, denatured and hybridised to the BeadChips for 20 h at 48 °C. The BeadChips were washed and the hybridised primers were extended and labelled before scanning the BeadChips using the Illumina iScan system. GenomeStudio software (version 2011.1; Illumina Inc.) was used for the extraction of DNA methylation signals from scanned arrays. The methylation level for each cytosine was expressed as a beta value calculated as the fluorescence intensity ratio of the methylated to unmethylated versions of the probes: beta values ranged between 0 (unmethylated) and 1 (methylated). The annotation relating to CGIs uses the following categorisation: 'shore', each of the 2-kb sequences flanking a CGI; 'shelf', each of the 2-kb sequences next to a shore; 'open sea', DNA not included in any of the previous sequences or in CGIs 4. TSS200 and TSS1500 indicate the region between position -200 bp and -1500 bp from the TSS, respectively. The significant methylation difference between two given loci is indicated by a delta-beta value and determined with GenomeStudio Methylation Module using Illumina custom algorithm for calculating DiffScores (DiffScore⩽-30.0 (≈ pval <0.001)=hypo-methylation; DiffScore⩾30.0 (≈ p val<0.001)=hyper-methylation).

ELIGIBILITY:
Inclusion Criteria for subjects with Episodic Migraine (EM):

1. satisfaction of the diagnostic criteria for migraine without aura according to the International Headache Classification 3rd edition (ICHD-3);
2. an episodic pattern of migraine for at least 10 years without any period of chronification.

Exclusion Criteria:

any systemic diseases, psychiatric disorders or any other clinically significant conditions.

Inclusion criteria for patient with chronic migraine with medication overuse (CM-MO):

1. satisfaction of the ICHD-3 diagnostic criteria for chronic migraine and for one of the subtypes of medication overuse headache;
2. a history of stable chronification for at least 5 years.

Exclusion Criteria:

any systemic diseases, psychiatric disorders or any other clinically significant conditions.

Inclusion Criteria for healthy controls (CT):

1. no history of migraine or other primary headaches;
2. Infrequent tension-type headache episodes.

Exclusion Criteria:

1. any systemic diseases, psychiatric disorders or any other clinically significant conditions;
2. any type of painkiller in the 24 hours prior to the blood sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with episodic migraine (EM), chronic migraine with medication overuse (CM-MO) and age-matched healthy controls (CT).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
CB1 (endocannabinoid receptor) protein expression | At the time of enrollment
  CB1 protein expression in the peripheral blood mononuclear cells (PBMCs)
CB2 (endocannabinoid receptor) protein expression | At the time of enrollment
  CB2 protein expression in the peripheral blood mononuclear cells (PBMCs)
Gene Expression of the CB receptors | At the time of enrollment
  Gene expression of the endocannabinoid receptors in the peripheral blood mononuclear cells ( PBMCs)
Gene Expression of the fatty acid amide hydrolase (FAAH) | At the time of enrollment
  Gene expression of the FAAH in the peripheral blood mononuclear cells ( PBMCs)
Gene Expression of the N-acylphosphatidylethanolamide-phospholipase D (NAPE-PLD) | At the time of enrollment
  Gene expression of the NAPE-PLD in the peripheral blood mononuclear cells ( PBMCs)
Gene Expression of the diacylglycerol lipase (DAGL) | At the time of enrollment
  Gene expression of the DAGL in the peripheral blood mononuclear cells ( PBMCs)
Gene Expression of the monoacylglycerol lipase (MAGL). | At the time of enrollment
  Gene expression of the MAGL in the peripheral blood mononuclear cells ( PBMCs)
DNA methylation of endocannabinoid system (ES) components | At the time of enrollment
  DNA methylation in the regulation of ES gene transcription

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, MD, Principal Investigator — IRCCS MONDINO FOUNDATION
Locations (1):
- Ircss Mondino Foundation, Pavia, Italy

REFERENCES:
- [Background] Basavarajappa BS, Nixon RA, Arancio O. Endocannabinoid system: emerging role from neurodevelopment to neurodegeneration. Mini Rev Med Chem. 2009 Apr;9(4):448-62. doi: 10.2174/138955709787847921. PMID 19356123
- [Background] Greco R, Demartini C, Zanaboni AM, Piomelli D, Tassorelli C. Endocannabinoid System and Migraine Pain: An Update. Front Neurosci. 2018 Mar 19;12:172. doi: 10.3389/fnins.2018.00172. eCollection 2018. PMID 29615860
- [Background] Greco R, Demartini C, Zanaboni AM, Tumelero E, Reggiani A, Misto A, Piomelli D, Tassorelli C. FAAH inhibition as a preventive treatment for migraine: A pre-clinical study. Neurobiol Dis. 2020 Feb;134:104624. doi: 10.1016/j.nbd.2019.104624. Epub 2019 Oct 17. PMID 31629892
- [Background] La Porta C, Bura SA, Llorente-Onaindia J, Pastor A, Navarrete F, Garcia-Gutierrez MS, De la Torre R, Manzanares J, Monfort J, Maldonado R. Role of the endocannabinoid system in the emotional manifestations of osteoarthritis pain. Pain. 2015 Oct;156(10):2001-2012. doi: 10.1097/j.pain.0000000000000260. PMID 26067584
- [Background] Centonze D, Battistini L, Maccarrone M. The endocannabinoid system in peripheral lymphocytes as a mirror of neuroinflammatory diseases. Curr Pharm Des. 2008;14(23):2370-42. doi: 10.2174/138161208785740018. PMID 18781987
- [Background] Sarchielli P, Pini LA, Coppola F, Rossi C, Baldi A, Mancini ML, Calabresi P. Endocannabinoids in chronic migraine: CSF findings suggest a system failure. Neuropsychopharmacology. 2007 Jun;32(6):1384-90. doi: 10.1038/sj.npp.1301246. Epub 2006 Nov 22. PMID 17119542
- [Background] Arosio B, Bulbarelli A, Bastias Candia S, Lonati E, Mastronardi L, Romualdi P, Candeletti S, Gussago C, Galimberti D, Scarpini E, Dell'Osso B, Altamura C, MacCarrone M, Bergamaschini L, D'Addario C, Mari D. Pin1 contribution to Alzheimer's disease: transcriptional and epigenetic mechanisms in patients with late-onset Alzheimer's disease. Neurodegener Dis. 2012;10(1-4):207-11. doi: 10.1159/000333799. Epub 2012 Jan 17. PMID 22261503
- [Background] Van der Schueren BJ, Van Laere K, Gerard N, Bormans G, De Hoon JN. Interictal type 1 cannabinoid receptor binding is increased in female migraine patients. Headache. 2012 Mar;52(3):433-40. doi: 10.1111/j.1526-4610.2011.02030.x. Epub 2011 Nov 11. PMID 22077199
- [Background] Perrotta A, Arce-Leal N, Tassorelli C, Gasperi V, Sances G, Blandini F, Serrao M, Bolla M, Pierelli F, Nappi G, Maccarrone M, Sandrini G. Acute reduction of anandamide-hydrolase (FAAH) activity is coupled with a reduction of nociceptive pathways facilitation in medication-overuse headache subjects after withdrawal treatment. Headache. 2012 Oct;52(9):1350-61. doi: 10.1111/j.1526-4610.2012.02170.x. Epub 2012 Jun 1. PMID 22670561
- [Background] Frieling H, Albrecht H, Jedtberg S, Gozner A, Lenz B, Wilhelm J, Hillemacher T, de Zwaan M, Kornhuber J, Bleich S. Elevated cannabinoid 1 receptor mRNA is linked to eating disorder related behavior and attitudes in females with eating disorders. Psychoneuroendocrinology. 2009 May;34(4):620-4. doi: 10.1016/j.psyneuen.2008.10.014. Epub 2008 Nov 28. PMID 19046818
- [Background] Greco R, Bandiera T, Mangione AS, Demartini C, Siani F, Nappi G, Sandrini G, Guijarro A, Armirotti A, Piomelli D, Tassorelli C. Effects of peripheral FAAH blockade on NTG-induced hyperalgesia--evaluation of URB937 in an animal model of migraine. Cephalalgia. 2015 Oct;35(12):1065-76. doi: 10.1177/0333102414566862. Epub 2015 Jan 21. PMID 25608877
- [Background] Greco R, Gasperi V, Sandrini G, Bagetta G, Nappi G, Maccarrone M, Tassorelli C. Alterations of the endocannabinoid system in an animal model of migraine: evaluation in cerebral areas of rat. Cephalalgia. 2010 Mar;30(3):296-302. doi: 10.1111/j.1468-2982.2009.01924.x. Epub 2010 Feb 1. PMID 19515121